CLINICAL TRIAL: NCT03698422
Title: Diurnal Variation in Markers of Mineral and Bone Disease in Chronic Kidney Disease - An Observational Study
Brief Title: Diurnal Variation in Markers of Mineral and Bone Disease in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ditte Hansen, Associate professor, Herlev Hospital
Other Study IDs: H-18037663
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Diseases; Mineral Metabolism Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma samples are collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Estimated glomerular filtration rate (eGFR) > 60 mL/min for > 3 months and no known current or chronic medical or surgical conditions.
  Blood and urine samples are collected for every 3rd hour during 24 hours
  Interventions: Diagnostic Test: Blood and urine samples
- Predialysis CKD subjects: Estimated glomerular filtration rate (eGFR) between 30 and 15 mL/min for > 3 months (i.e. CKD stage 4).
  Blood and urine samples are collected for every 3rd hour during 24 hours
  Interventions: Diagnostic Test: Blood and urine samples
- ESKD subjects: Maintenance haemodialysis treatment for > 3 months for ESKD and with anuria (urine excretion < 100 mL/day).
  Blood and urine samples are collected for every 3rd hour during 24 hours
  Interventions: Diagnostic Test: Blood and urine samples

INTERVENTIONS:
Diagnostic Test: Blood and urine samples — Subjects will be admitted to the Department of Nephrology, Herlev and Gentofte Hospital, Herlev, Denmark, for 24-hour observation with measurements of serum and urine at three-hour intervals.

SUMMARY:
The purpose of this study is to examine whether there are diurnal variations in magnesium and other markers related to mineral metabolism in blood from patients with chronic kidney disease (CKD) compared to healthy controls.

DETAILED DESCRIPTION:
CKD is associated with a mortality rate 5-10 times higher than in the general population, which is driven by a high rate of cardiovascular disease. Several cohort studies have revealed an association between hypomagnesaemia and increased mortality in patients with CKD as well as faster progression of CKD. Additionally, studies in cultured vascular smooth muscle cells (VSMC) and in rodents with CKD have shown that Mg inhibits vascular calcification.

The exact mechanism behind the inhibitory effect of Mg on vascular calcification is incompletely understood, but seems to be related to an inhibitory effect on the formation and precipitation of hydroxyapatite and delayed formation of secondary calciprotein particles, both of which have been shown to induce calcification of VSMC in vitro. Mg blocks the calcium (Ca) influx across the cell membrane in the VSMC. Mg has some affinity for the Ca sensing receptor, which has been shown to be involved in the calcification of VSMC, and might thus inhibit vascular calcification in a manner similar to other calcimimetics.

Thus, increasing serum Mg has been proposed as a possible treatment to prevent vascular calcification in CKD. However, any diurnal variation in serum Mg and other markers of mineral metabolism related to vascular calcification in CKD have not previously been described. This is relevant as monitoring of treatment with Mg supplementation might potentially be dangerous, if there are significant diurnal changes in serum Mg. Therefore, we wish to conduct a prospective controlled clinical trial to investigate any diurnal changes in Mg other markers of mineral metabolism in healthy controls, patients with predialysis CKD and patients with end-stage kidney disease (ESKD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Serum Mg between 0.7 and 1.1 mmol/L on average of previous measurements over the last 6 months.
* Serum ionised Ca between 1.10 and 1.35 mmol/L on average of previous measurements over the last 6 months.
* Serum phosphate (PO4) between 0.7 and 1.8 mmol/L on average of previous measurements over the last 6 months.
* A negative pregnancy test for women of childbearing age.
* Written informed consent.
* For healthy controls - estimated glomerular filtration rate (eGFR) > 60 mL/min for > 3 months and no known current or chronic medical or surgical conditions.
* For predialysis CKD subjects - estimated glomerular filtration rate (eGFR) between 30 and 15 mL/min for > 3 months (i.e. CKD stage 4).
* For ESKD subjects - maintenance haemodialysis treatment for > 3 months for ESKD and with anuria (urine excretion < 100 mL/day).

Exclusion Criteria:

* Diagnosis of diabetes mellitus.
* Kidney transplant recipient.
* Parathyroid hormone (PTH) > 66 ρmol/L during the previous 3 months.
* Previous parathyroidectomy.
* Current treatment with Mg containing medication or supplements.
* Current treatment with calcimimetics.
* Current treatment with immunosuppressive drugs.
* Active malignant disease.
* Blood haemoglobin < 6.0 mmol/L
* Any condition impairing Mg absorption from the gastrointestinal tract (e.g. short bowel syndrome, chronic pancreatitis).
* Other diseases or conditions, which, in the opinion of the site investigator, would prevent participation in or completion of trial.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For healthy controls:
  estimated glomerular filtration rate (eGFR) > 60 mL/min for > 3 months and no known current or chronic medical or surgical conditions.
  For predialysis CKD subjects:
  estimated glomerular filtration rate (eGFR) between 30 and 15 mL/min for > 3 months (i.e. CKD stage 4).
  For ESKD subjects:
  maintenance haemodialysis treatment for > 3 months for ESKD and with anuria (urine excretion < 100 mL/day).
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Diurnal change in serum magnesium within groups | 24 hours
  change in serum magnesium (mmol/l) within Groups The changes within groups over several timepoints will be compared with linear mixed effect models

SECONDARY OUTCOMES:
Change in serum magnesium between groups | 24 hours
  Change in serum magnesium (mmol/l) between Groups The overall magnesium levels will be compared between groups by comparing the total mean of measurements for each group.
Change in ionized calcium | 24 hours
  Change in p-ionized calcium within and between groups
Change in p-phosphate | 24 hours
  Change in p-phosphate within and between groups
Change in p-PTH | 24 hours
  Change in p-PTH within and between groups
Change in p-FGF23 | 24 hours
  Change in p-FGF23 within and between groups
Change in s-calcification propensity score | 24 hours
  Change in s-calcification propensity score within and between groups
Change in u-magnesium | 24 hours
  Change in u-magnesium within and between groups

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, PhD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No